CLINICAL TRIAL: NCT02561234
Title: A Multiple Dose, Dose Escalation Trial of AEB1102 (Co-ArgI-PEG) in Patients With Advanced Solid Tumors
Brief Title: A Multiple Dose, Dose Escalation Trial of AEB1102 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aeglea Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAEB1102-100B
Record Dates: First submitted 2015-08-25; First posted 2015-09-28 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Advanced Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- AEB1102 Dose Escalation Cohort 1 (Experimental): 3 patients dosed at 0.01 mg/kg until MTD determined
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Dose Escalation Cohort 2 (Experimental): 4 patients dosed at 0.02 mg/kg until MTD determined
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Dose Escalation Cohort 3 (Experimental): 4 patients dosed at 0.04 mg/kg until MTD determined
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Dose Escalation Cohort 4 (Experimental): 4 patients dosed at 0.08 mg/kg until MTD determined
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Dose Escalation Cohort 5 (Experimental): 3 patients dosed at 0.12 mg/kg until MTD determined
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Dose Escalation Cohort 6 (Experimental): 4 patients dosed at 0.18 mg/kg until MTD determined
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Dose Escalation Cohort 7 (Experimental): 5 patients dosed at 0.27 mg/kg until MTD determined
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Dose Escalation Cohort 8 (Experimental): 7 patients dosed at 0.40 mg/kg until MTD determined
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Dose Escalation Cohort 9 (Experimental): 7 patients dosed at 0.33 mg/kg until MTD determined MTD determined at 0.33 mg/kg
  Interventions: Drug: Co-ArgI-PEG
- AEB1102 Expansion (Experimental): Uveal: 11 patients dosed at 0.33 mg/kg Cutaneous Melanoma: 11 dosed at 0.33 mg/kg SCLC: 13 patients dosed at 0.33 mg/kg
  Interventions: Drug: Co-ArgI-PEG

INTERVENTIONS:
Drug: Co-ArgI-PEG — Administered IV
  Other Names: AEB1102

SUMMARY:
This is the first-in-human study of the safety of increasing dose levels of AEB1102 in patients with advanced cancers. The study will also evaluate the amounts of AEB1102 in blood, the effects of AEB1102 on blood amino acid levels and tumor growth.

DETAILED DESCRIPTION:
In this phase I/2 multiple dose, dose escalation study utilizing a classic 3+3 design. Sequential cohorts of patients will receive AEB1102 IV weekly at one of a series of increasing dose levels. Dose escalation will be dependent on the frequency of specific dose-limiting toxicities in the prior cohort of patients. The study will determine the maximum tolerated dose (MTD) of AEB1102, evaluate the safety profile of the compound, assess the pharmacokinetic profile of AEB1102, determine the effect of AEB1102 on blood arginine levels and evaluate the anti-tumor activity of AEB1102.

Following the determination of the MTD, additional cohorts of patients with uveal, cutaneous melanoma and small cell lung cancer will be enrolled and treated with AEB1102 at the MTD.

ELIGIBILITY:
Inclusion Criteria:

For patients participating in any part of the trial:

* has an advanced solid tumor previously treated with, or inability to tolerate, standard therapy for the disease, or for which a standard therapy does not exist, and as such is considered a candidate for Phase 1 treatment
* has adequate organ function: Hgb ≥9 g/dL; absolute neutrophil count (ANC) ≥ 1.5x109/L; plt ≥ 100,000/μL; AST and ALT < 2.5x ULN (< 5x ULN in patients with liver metastases); total bilirubin < 2.0 mg/dL; serum creatinine ≤ 1.5x ULN
* ECOG performance score 0-2

For patients participating in any expansion group:

* has measurable disease based on RECIST 1.1 as determined by the treating investigator. Tumor lesions in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* willing to consent for biopsy is strongly recommended but not mandatory
* recovery of toxicities related to any prior treatments to at least Grade 1 by CTCAE v 4.03. Exceptions are patients with adverse event(s) that are clinically nonsignificant and/or stable on supportive therapy.

For patients participating in specific expansion groups:

Cutaneous Melanoma:

* unresectable, locally advanced or metastatic (AJCC stage IIIB, IIIC, or IV) cutaneous malignant melanoma
* relapsed or progressive disease after or unable to tolerate at least one prior systemic anticancer regimen for metastatic disease involving immunotherapy (anti-PD-1, anti-PD-L1, or anti-CTLA-4)
* in tumors with a relevant BRAF mutation, relapsed, refactory, or unable to tolerate at least one prior systemic anticancer regimen for metastic disease involving a BRAF inhibitor

Uveal Melanoma:

* uveal melanoma at metastic stage

Small Cell Lung Cancer:

* extensive disease previously treated with, or inability to tolerate, platinum-based chemotherapy

Exclusion Criteria:

* has primary CNS malignancy
* history of untreated brain mets or leptomeningeal disease or spinal cord compression
* effects of prior anticancer therapy recovered to grade < 2
* known HIV
* active infection
* major surgery within 2 weeks
* history of another malignancy within 2 years prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-10; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 4 weeks
  the dose level at which no more than 1/6 patients experiences dose-limiting toxicity

SECONDARY OUTCOMES:
safety profile (changes in physical exam, laboratory measures, reported adverse events) | 4 weeks +
  changes in physical exam, laboratory measures, reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jim Joffrion, Study Director — Aeglea Biotherapeutics, Inc.
Locations (11):
- United States (11):
  - Pinnacle Research, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Research Center: Mid Florida Hematology/Oncology Centers, Orange City, Florida
  - Dana Farber, Boston, Massachusetts
  - Massachusetts General, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Providence Cancer Center, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UTSW, Dallas, Texas